CLINICAL TRIAL: NCT06045871
Title: Evaluation of Surgical Correction of Anterior Vertical Maxillary Excess (Gummy Smile) by Compression.
Brief Title: Evaluation of Surgical Correction of Anterior Vertical Maxillary Excess (Gummy Smile) by Compression Osteogenesis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Samir El-helaly, Principal investigator., Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OMFS 3.3.2
Record Dates: First submitted 2023-09-04; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Compression Osteogenesis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with anterior vertical maxillary excess (gummy smile) (Other)
  Interventions: Procedure: Corticotomy followed by compression osteogenesis

INTERVENTIONS:
Procedure: Corticotomy followed by compression osteogenesis — Surgical corticotomy supra apical in anterior maxilla then application of the compression osteogenesis concept via traction on miniscrews implanted above the corticotomy line

SUMMARY:
The technique of compression osteogenesis will be studied to verify its value as applied to manage anterior vertical maxillary excess in patients wohm are suffering from gummy smile.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from anterior vertical maxillary excess that requires surgical intervention

Exclusion Criteria:

* total vertical maxillary excess Excessive horizontal maxillary excess Patients with systemic diseases that may affect normal bone healing

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2023-02-02 (Actual)

PRIMARY OUTCOMES:
Measuring amount of vertical impaction of anterior maxilla after performing labial maxillary cotricotomy and activation of functional loading | 3 months
  Measuring amount of linear impaction (in millimeters) to evaluate validity of compression osteogenesis in treating gummy smile of a skeletal etiology ( due to increased anterior maxilla height) after performing labia maxillary corticotomy and activating functional loading using power chain elastics anchored on transmucosal mini- screws.

CONTACTS AND LOCATIONS:
Locations (1):
- Marwa Elhelaly, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes